CLINICAL TRIAL: NCT01209039
Title: A Healthy Volunteer Repeat Dose Study to Evaluate; the Safety, Tolerability, Pharmacokinetics, Effects on the Pharmacokinetics of Midazolam and the Neurokinin 1 Receptor Occupancy of GSK1144814
Brief Title: A Repeat Dose Positron Emission Tomography Study With GSK1144814
Acronym: NK1 NK3 PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 111587
Record Dates: First submitted 2010-08-30; First posted 2010-09-24 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; PET
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part A, cohort 1 and 2 (Experimental): Part A, Cohorts 1 and 2, will investigate escalating multiple daily doses of GSK1144814 in 19 subjects
  Interventions: Drug: GSK1144814
- Part A, cohort 3 (Experimental): Cohort 3 will investigate safety, tolerability and PK of a dose of GSK1144814 over a repeat treatment period of 28 days in 18 subjects and a potential drug drug interaction between GSK1144814 and the CYP3A4 sensitive substrate midazolam (in 15 subjects).
  Interventions: Drug: GSK1144814
- Part B (Experimental): Part B will assess NK1 receptor occupancy following repeated administration of GSK1144814 given once daily until steady state is obtained
  Interventions: Drug: GSK1144814

INTERVENTIONS:
Drug: GSK1144814 — Multiple daily doses of GSK1144814 for 28 days
  Arms: Part A, cohort 3
Drug: GSK1144814 — Multiple daily doses of GSK1144814 for 14 days
  Arms: Part A, cohort 1 and 2
Drug: GSK1144814 — Multiple daily doses of GSK1144814 for 7 days (or until steady state is reached)
  Arms: Part B

SUMMARY:
This study described in the present protocol consists of two parts. Part A is a multiple ascending dose study to evaluate the safety, tolerability and pharmacokinetics of ascending doses of GSK1144814. Part B is an open label design in healthy male subjects to assess the GSK1144814 Neurokinin1 receptor occupancy.

DETAILED DESCRIPTION:
GSK1144814 is a dual Neurokinin 1 and Neurokinin 3 antagonist with the potential to treat schizophrenia and depression.

This study described in the present protocol consists of two parts. Part A is a multiple ascending dose study to evaluate the safety, tolerability and pharmacokinetics of ascending doses of GSK1144814. The study is a single blind, randomised, placebo controlled design in healthy male and female (of non childbearing potential) subjects. Part B is an open label design in healthy male subjects to assess the GSK1144814 Neurokinin 1 receptor occupancy after repeat oral dosing by positron emission tomography scanning with [11C] GR205171.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if, in the opinion of the Investigator, the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female aged between 18 and 65 years (inclusive) for Part A, or male aged between 25 and 55 years (inclusive) for Part B.
* A female subject is eligible to participate in Part A if she is of:

Non childbearing potential defined as pre menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] higher than 40 mIU/mL and oestradiol lower than 40 pg/mL [lower than 140 pmol/L] is confirmatory).

* Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to discontinue HRT to allow confirmation of post menopausal status prior to study enrolment. For most forms of HRT, at least 2 to 4 weeks will elapse between the cessation of therapy and the blood sampling; this interval depends on the type and dosage of HRT. Following confirmation of their post menopausal status, they can resume the use of HRT during the study without the use of a contraceptive method.
* A male subject must agree to use one of the contraception methods listed in Section 8.1.2. This criterion must be followed from the first investigational product dosing day until at least 3 months after receiving the last dose of the investigational product.
* Body weight higher than or equal to 50 kg and body mass index (BMI) within the range 18 to 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTcB or QTcF lower than 450 msec.
* Demonstrates no evidence of mental impairment or co morbid psychiatric disorders or suicidal risk (as determined with the Columbia Suicide Severity Rating Scale [C SSRS]).

Exclusion Criteria:

* The subject has a positive pre study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre study hepatitis B surface antigen (HBsAg) or positive hepatitis C virus (HCV) antibody test result within 3 months of Screening.
* A positive test result for antibodies to human immunodeficiency virus (HIV) 1/2.
* Significant renal abnormality (from medical history or as indicated by laboratory investigations. In addition, subjects with idiopathic haematuria or proteinuria or conditions such as benign orthostatic proteinuria and benign familial haematuria should be excluded from the study).
* History of regular alcohol consumption within 6 months of the study start defined as:

An average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half pint (220 mL) of beer or 1 measure (25 mL) of spirits or 1 glass (125 mL) of wine.

* The subject has participated in a clinical trial and has received an investigational product within 3 month prior to the first investigational product dosing day in the current study.
* Exposure to more than four new chemical entities within 12 months prior to the first investigational product dosing day.
* Use of prescription or non prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half lives (whichever is longer) prior to receiving the first dose of the investigational product, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the investigational products, or components thereof or a history of drug or other allergy that, in the opinion of the Investigator or GSK Medical Monitor, contraindicates their participation in the study.
* Where participation in the study would result in donation of blood or blood products in excess of 600 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* History or presence of clinically significant cardiac arrhythmias, or other clinically significant cardiac disease.
* Smokers confirmed by a positive urinary cotinine test (greater than the local laboratory lower limit of quantification [LLQ] of 200 ng/mL or lower). Urine cotinine levels will be measured during Screening and at Baseline.
* Consumption of Seville oranges (including marmalade) and/or grapefruit and/or Chinese grapefruit (pomelo) and/or grapefruit hybrids and/or exotic citrus fruits and/or their fruit juices from 7 days prior to the first investigational product dosing day.
* Consumption of red wine from 7 days prior to the first investigational product dosing day.

For Part B only:

* Abnormal Allen's test for adequate collateral blood flow to the hand.
* Previous inclusion in a research and/or medical protocol involving nuclear medicine, PET or radiological investigations with significant radiation burden (a significant radiation burden being defined as International Commission on Radiological Protection (ICRP) Category IIb or above: No more than 10 mSv in addition to natural background radiation, in the previous 3 years including the dose from this study).
* Family history of cancer (one or more first degree relative diagnosed before the age of 55 years, inclusive).
* History of or suffers from claustrophobia or feels that they will be unable to lie still on their back in the PET camera for a period of approximately 2 hours.
* History of neurological or psychiatric conditions (e.g., stroke, traumatic brain injury, epilepsy, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischaemic attack, schizophrenia, major depression, etc) that may influence the outcome or analysis of the scan results.
* Presence of a cardiac pacemaker or other electronic device or ferromagnetic metal foreign bodies in vulnerable positions as assessed by a standard pre MRI questionnaire supported by plain X rays where appropriate.
* Abnormal blood clotting profile, i.e., prolonged prothrombin time (INR).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-07-01 (Actual); Primary Completion 2009-10-25 (Actual); Study Completion 2009-10-25 (Actual)

PRIMARY OUTCOMES:
PET receptor occupancy | 1 week
To assess the safety and tolerability by reviewing the number of subjects with adverse events, a review of laboratory samples and a review of vitals. | 2 or 4 weeks
To review pharmacokinetic data | 2 or 4 weeks

SECONDARY OUTCOMES:
To assess potential induction of CYP3A4 | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United Kingdom (2):
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, London

REFERENCES:
- See also: Results for study 111587 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/111587?search=study&search_terms=111587#rs